CLINICAL TRIAL: NCT02531620
Title: Prehabilitation Interventions in Elective Colorectal Resections: A Randomized Pilot Study (Prehab)
Brief Title: Prehabilitation in Elective Colorectal Resection: A Pilot Study (Prehab)
Acronym: Prehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015A1
Record Dates: First submitted 2015-08-19; First posted 2015-08-24 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
Keywords: prehabilitation; colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiatry (Experimental): Pre-operative Physiatry assessment and intervention
  Interventions: Other: Physiatry Assessment
- Routine Care (Other): Patients will receive routine pre-operative care, this study arm does not have an intervention.
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Physiatry Assessment — Physiatrists are physicians who are medical experts in maximizing a patient's overall ability to function well and live independently. The Investigators are proposing your participation in an initial pilot study in order to test the question as to whether or not participation with a physiatrist and any interventions recommended by said physician would help improve a patient's postoperative recovery.
  Arms: Physiatry
Other: Routine Care — Usual care for your disease process
  Other Names: Standard Care
  Arms: Routine Care

SUMMARY:
This is a pilot study designed to evaluate a programme of rehabilitation for patients undergoing elective colorectal resection surgery.

DETAILED DESCRIPTION:
Operations on the colon and rectum are major abdominal operations and many individuals can become severely deconditioned or weakened afterwards. For some individuals this can even mean that they can no longer completely return to their usual way of life following one of these major operations. As part of this study the investigators are attempting to identify ways to maximize patients' recovery and to maximize their overall quality of life following these major operations. It is possible that preconditioning may make a difference to patient's overall quality of life, decreased or need for hospital length of stay and decreased postoperative medical complications occasionally seen during these operations, in essence provide an overall enhancement to their surgical recovery. Physiatrists are physicians who are medical experts in maximizing a patient's overall ability to function well and live independently. Investigators are proposing patient participation in an initial pilot study in order to test the question as to whether or not participation with a physiatrist and any interventions recommended by said physician would help improve a patient's postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* scheduled to undergo a colorectal resection as part of treatment for colorectal cancer.
* English speaking or have available a family member or substitute decision maker who can accompany you to all of your study visits.

Exclusion Criteria:

* geographic inaccessibility
* unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruiting | 6 months
  Screening and recruiting of eligible patients

SECONDARY OUTCOMES:
Post-op complications | 30 days
  Post-op complications by Clavien-Dindo classification (pulmonary, DVT, MI) Completed by surgical team during admission, discharge and 30 days
Mortality | 6 months
  Survival will be noted at completion of 6 month study period.
Length of Stay | 30 days post-op
  Length of stay in hospital will be collected and compared for the two treatment groups
Number of patients with readmissions | 30 days and 6 months
  Number of patients with readmission to hospital during the 30 day and 6 month period will be compared for the two treatment groups
Physical Function Assessment (6 Minute Walk Test) | 1, 3 and 6 months
  6 Minute Walk Test (6MWT)
Symptom Assessment (Edmonton Symptom Assessment System) | 1, 3 and 6 months
  Edmonton Symptom Assessment System (ESAS)
Functional Independence Assessment (UK Functional Independence Measure and Functional Assessment Measure) | 1, 3 and 6 months
  UK Functional Independence Measure and Functional Assessment Measure (UK FIM+FAM)
Quality of Life Survey (Short Form 36 Health Survey) | 1, 3 and 6 months
  Short Form 36 Health Survey (SF-36)
Pain Assessment (Visual Analog Scale) | 1, 3 and 6 months
  Pain score by Visual Analog Scale
Bowel Function Assessment | 1, 3 and 6 months
  Bowel Function Index

CONTACTS AND LOCATIONS:
Overall Officials: Nalin Amin, MD, Principal Investigator — McMaster University
Locations (1):
- St Joseph Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong SG, Maida E, Harvey D, Wagner N, Sonnadara R, Amin N. Evaluation of a physiatrist-directed prehabilitation intervention in frail patients with colorectal cancer: a randomised pilot study protocol. BMJ Open. 2017 Jun 9;7(6):e015565. doi: 10.1136/bmjopen-2016-015565. PMID 28600373